CLINICAL TRIAL: NCT01817283
Title: Study of Triptolide Woldifiion T Cell Immune Activation and Inflammation Biomarkers in HIV-infected Immunological Non-responders
Brief Title: Impact on T Cell Immune Activation and Inflammation of Triptolide Woldifii in HIV-infected Immunological Non-responders
Acronym: CACTrip12
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LI Taisheng (Other)
Responsible Party: Sponsor-Investigator, LI Taisheng, Peking Union Medical College Hospital, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CACTRIP12
Record Dates: First submitted 2013-03-18; First posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: HIV
Keywords: HIV-infected immunological non-responders; Triptolide; immune activation; inflammation; CD4 T cell
MeSH Terms: conditions — Inflammation | interventions — triptolide; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo + cART (Placebo Comparator): combined with antiretroviral therapy, the control group will take placebo 2 tabs tid per day lasting for 6 months and then switch to take Triplitode 2 tabs tid po for anther 6 months
  Interventions: Drug: Triptolide; Drug: cART; Drug: placebo
- Triptolide + cART (Experimental): combined antiretroviral therapy, the experimental group will take Triptolide 2 tabs tid po per day for 12 months.
  Interventions: Drug: Triptolide; Drug: cART

INTERVENTIONS:
Drug: Triptolide — Triptolide Wilfordii is a Chinese old herb which is widely used as a remedy for rheumatic diseases and nephropathy in China. It is approved that it can play a role as an immune modular.
  Other Names: Tripterygium Wilfordii Hook F (TwHF)
Drug: cART — Participants who will be enrolled in this trial would keep their previous combined antiretroviral therapy, such as zidovudine or stavudine plus lamivudine plus nevirapine or efavirenz.
  Other Names: Antiretroviral therapy
Drug: placebo — Placebo pills produced the same as Triptolide wilfordii.
  Other Names: sugar pills
  Arms: placebo + cART

SUMMARY:
This study is a prospective, multicenter, randomized, placebo-controlled clinical trial, to evaluate impact of Triptolide wilfordii on T cell immune activation and inflammation biomarkers in HIV-infected immunological non-responders.

DETAILED DESCRIPTION:
About 120 patients will be recruited from 4 HIV/AIDS clinical centers in China and randomized 1:1 into intervention group and placebo-controlled group. Triptolide wilfordii (20mg tid po) would be given to invention group for 24 weeks. T cell activation and inflammation biomarkers including CD8+HLA-DR+CD38+, IL-6, D-Dimer and high-sensitivity C-reactive protein (hsCRP), protein degradation-1 (PD-1), Ki67 ,soluble CD14 and CD163, PD-1, CCR5 and CD57 would be tested. Patients in placebo-controlled group will change to take Triptolide wilfordii (20mg tid po) for another 24 weeks. All patients will be followed up till 48 weeks. We hypothesis that Triptolide wilfordii might reduce immune activation and inflammation of HIV immunological non-responders and increase CD4 T cell count, which provides a new strategy for treatment of HIV-infected immunological non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Continuous antiretroviral therapy > 24 months ， and consistent HIV-RNA< 40 copies/mL more than 12 months ;
* 18-65 years old;
* Male or female;
* Good adherence and promise to follow-up;
* Inform Consent signed;
* CD4 T cells less than 250/ul .

Exclusion Criteria:

* Active opportunistic infection (not stable within 4 weeks 2 weeks ) or AIDS-related carcinoma;
* hemoglobin (HGB) < 9 g/dl 、 white blood cell (WBC) < 2000/ul 、 granulin (GRN) < 1000 /ul 、 platelet (PLT) < 75000 /ul 、 Cr >1.5x ULN 、 ALT or AST or alkaline phosphatase (ALP) >3x upper limit of normal (ULN) 、 total bilirubin (TBIL) >2x ULN 、 creatine kinase (CK) > 2x ULN;
* Pregnant or breastfeeding woman or woman with pregnancy plan;
* Active drug-user;
* Severe neurological defects;
* Active alcohol abuse;
* Severe gastrointestinal ulcer .
* End-stage disease such as cirrhosis, chronic obstructive pulmonary disease, congestive heart failure, recent myocardial ischemia,tumor, etc
* Those who are undertaking steroids, immunomodulator, anti-inflammatory agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Changes of T cell immune activation and inflammation biomarkers | baseline and at 4,8,12,24,36,48 weeks
  T cell activation and inflammatory biomarkers including CD8+HLA-DR+/CD38+, IL-6, D-dimer and hsCRP,soluble CD14 and CD163, PD-1, CCR5 and CD57 should be measured at baseline and at Wee4, W12, W24, W36, W48 follow-up visits.

SECONDARY OUTCOMES:
Changes of CD4 T cell count and number of participants with adverse events | baseline and at 4,8,12,24,36,48 weeks
  Measurement of CD4 T cell count at baseline and different visit points when follow-up and numbers of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Tai sheng LI, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China